CLINICAL TRIAL: NCT06296576
Title: Acceleration Time Assessment for Prediction of Critical Limb Ischemia
Acronym: ATACLI
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier le Mans (Other)
Responsible Party: Sponsor
Other Study IDs: CHM-2023/S49/06
Record Dates: First submitted 2024-02-29; First posted 2024-03-06 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-02

CONDITIONS: Critical Limb Ischemia
Keywords: systolic rise time; critical limb ischaemia
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: arterial ultrasound scan — An arterial ultrasound scan of the lower limbs with pulsed Doppler analysis of arterial flow spectra over the abdominal aorta, dorsal artery of the foot and lateral plantar artery, bilaterally

SUMMARY:
Critical Limb Ischaemia (CLI), the final stage of arterial disease, is a therapeutic emergency whose prognosis depends largely on the time taken to diagnose it. The growing prevalence of this condition and the associated healthcare costs make it an important public health objective. Diagnostic criteria for Critical Limb Ischaemia differ between learned societies and countries.

Its diagnosis is most frequently based on the combination of a clinical criterion (ischaemic decubitus pain and/or necrotic wounds, with a time to onset > 2 weeks) and a haemodynamic criterion (ankle systolic pressure (ASP) < 50mmHg or toe systolic pressure (TSP) < 30 mmHg or transcutaneous oxygen pressure (TCPO2) < 30 mmHg).

Recent studies have highlighted the importance of pulsed Doppler flow analysis in quantifying arteriopathy of the lower limbs, both by systematically analysing flow modulation and by measuring the systolic rise time of distal arteries (dorsal artery of the foot and lateral plantar artery).

The main aim of this study is therefore to validate a reliable and accessible diagnostic tool for screening patients suffering from CLI so that they can be referred to a reference centre as early as possible.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* Patient referred to the vascular medicine department of one of the investigating centres for arterial Doppler ultrasound of at least one lower limb and for whom a measurement of the systolic pressure index at the toe will be performed.
* Presence of proven arterial disease, asymptomatic or not, defined by the presence of one of the following criteria:

  * Rest ankle systolic pressure index ≤ 0.90
  * Rest toe systolic pressure index ≤ 0.70

Exclusion Criteria:

* Patient with haemodynamic instability, unable to tolerate a delay in therapeutic management caused by the ultrasound examination and measurement of systolic pressure at the toe;
* Patients with surgical management of the lower limb (in relation to lower limb arteriopathy), already scheduled at the time of inclusion.
* Patients with a life expectancy of less than 24 hours;
* History of transmetatarsal amputation or amputation at a more proximal level compromising the measurement of systolic pressure and occlusion at the toe and/or TCPO2;
* Refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient referred to the vascular medicine department of one of the investigating centres for arterial Doppler ultrasound of at least one lower limb
Sampling Method: Non-Probability Sample
Enrollment: 431 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate the intrinsic diagnostic performance of the maximum systolic rise time (TASmax) in the distal arteries of the foot | 12 months
  The diagnosis of Critical Limb ischaemia will be defined by a toe systolic pressure ≤ 30 mmHg

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Centre Hospitalier de CHOLET, Cholet
  - Centre Hospitalier du Mans, Le Mans
  - CHU Poitiers, Poitiers